CLINICAL TRIAL: NCT02528682
Title: Vaccination With PD-L1/L2-silenced Minor Histocompatibility Antigen-loaded Donor DC Vaccines to Boost Graft-versus-tumor Immunity After Allogeneic Stem Cell Transplantation (a Phase I/II Study)
Brief Title: MiHA-loaded PD-L-silenced DC Vaccination After Allogeneic SCT
Acronym: PSCT19
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Dutch Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSCT19
Record Dates: First submitted 2015-08-18; First posted 2015-08-19 (Estimated); Last update posted 2021-04-01 (Actual); Status verified 2021-01

CONDITIONS: Hematological Malignancies
Keywords: dendritic cells; PD-L1/L2 silencing; vaccination; stem cell transplantation; minor histocompatibility antigens
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental): MiHA-loaded PD-L-silenced DC Vaccination
  Interventions: Biological: MiHA-loaded PD-L-silenced DC Vaccination

INTERVENTIONS:
Biological: MiHA-loaded PD-L-silenced DC Vaccination — Eligible patients will receive one cycle of donor DC vaccination consisting of maximal 3 immunizations, given at 2 week intervals. PD-L1/L2-silenced, MiHA mRNA-electroporated donor DC will be infused intravenously (2.5x105/kg body weight).

SUMMARY:
Allogeneic stem cell transplantation (allo-SCT) is a potent treatment, and sometimes the only curative treatment for aggressive hematological malignancies. The therapeutic efficacy is attributed to the graft-versus-tumor (GVT) response, during which donor-derived CD8+ T cells become activated by recipient minor histocompatibility antigens (MiHA) presented on dendritic cells (DC). Consequently, these alloreactive donor T cells clonally expand, acquire effector functions and kill MiHA-positive malignant cells. However, in a substantial number of patients persistence and recurrence of malignant disease is observed, indicating that insufficient GVT immunity is induced. This is reflected by our observation that not all patients develop a productive CD8+ T cell response towards MiHA mismatched between the recipient and donor. We found that the PD-1/PD-L1 co-inhibitory pathway is involved in dampening MiHA-specific CD8+ T cell expansion and function post-transplantation. Therefore, a promising strategy to induce or boost GVT immune responses is pre-emptive or therapeutic vaccination with ex vivo-generated donor DCs loaded with MiHA that are exclusively expressed by recipient hematopoietic cells and their malignant counterparts. In contrast to pre-emptive donor lymphocyte infusion (DLI) with polyclonal donor T cells, this MiHA-DC vaccination approach has less risk of inducing graft-versus-host disease (GVHD) and the potency to induce more efficient GVT-associated T cell immunity. In addition, the potency of this DC vaccine will be further enhanced by interference with the PD-1/PD-L1 co-inhibitory pathway, using siRNA mediated PD-L1/PD-L2 silencing.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AML, myelodysplasia (MDS), ALL, CML (accelerated or blast phase), CLL, MM, malignant NHL or HL, who underwent HLA-matched allo-SCT
* Patients positive for HLA-A2 and/or HLA-B7
* Patients positive for HA-1, LRH-1 and/or ARHGDIB transplanted with corresponding MiHA-negative donor
* Patients ≥18 years of age
* WHO performance 0-2
* Witnessed written informed consent

Exclusion Criteria:

* Life expectancy < 3 months
* Severe neurological or psychiatric disease
* Progressive disease needing cytoreductive therapy
* HIV positivity
* Patients with acute GVHD grade 3 or 4
* Patients with severe chronic GVHD
* Patients with active infections (viral, bacterial or fungal) that require specific therapy. Acute anti-infectious therapy must have been completed within 14 days prior to study treatment
* Severe cardiovascular disease (arrhythmias requiring chronic treatment, congestive heart failure or symptomatic ischemic heart disease)
* Severe pulmonary dysfunction
* Severe renal dysfunction (serum creatinine > 3 times normal level)
* Severe hepatic dysfunction (serum bilirubin or transaminases > 3 times normal level)
* Patients with known allergy to shell fish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-01; Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of toxicity | From day 0 until day 84
  Toxicity will be measured using the NCI CTCAE criteria (http://ctep.cancer.gov/reporting/ctc.html). Possible toxicities include constitutional symptoms such as fever, chills, myalgias, malaise and allergic reactions.
Development of GVHD | From day 0 until day 84
  DC vaccination may result in GVHD, which will be scored and treated if indicated according to standard guidelines.
The generation and magnitude of an immunological response | From day 0 until day 84
  When after DC vaccination >1.0% of all CD8+ lymphocytes at any time point are specific CD8+ T cells to the used MiHA vaccine target, a complete response will be considered to be present. When the percentage is between 0.02% and 1%, but has been doubled during two weeks, a partial immune response will be considered to be present.

SECONDARY OUTCOMES:
Changes in chimerism | day 0, day 14, day 28, day 64, day 84
  When chimerism changes towards donor or disease load decreases according to objective standard clinical criteria after vaccination, this will be considered as a clinical response.
  Chimerism in PBMC will be measured by SNP Q-PCR analysis according to standard practice in the molecular diagnostic unit of Department of Laboratory Medicine. When chimerism changes towards complete donor, this will be considered as a clinical response.
Disappearance of residual disease | day 0, day 14, day 28, day 64, day 84
  In the case of presence of detectable residual or persistent disease before DC vaccination, clinical effects will be investigated by monitoring residual disease by quantitative real-time bcr-abl PCR (CML, Ph+ ALL), WT1-specific PCR (AML, MDS), M-protein (MM), immunophenotyping (CLL, AML, ALL, MDS) and radiological examination (NHL) after vaccination. When disease load decreases according to objective standard clinical criteria after vaccination, this will be considered as a clinical response.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas Schaap, MD/PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Trialoffice Haematology-Oncology, Nijmegen, Gelderland, Netherlands